CLINICAL TRIAL: NCT02972320
Title: Lobaplatin Combined With Etoposide for First-line Treatment in Extensive Stage Sclc Then Benefit Patients Follow up Temozolomide Maintain Therapeutic
Brief Title: Extensive Stage Sclc Patients Who Were Benefit From First-line Treatment Accept Temozolomide Maintain Therapeutic
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yunpeng Liu (Other)
Responsible Party: Sponsor-Investigator, Yunpeng Liu, Director, clinical research, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOG1601
Record Dates: First submitted 2016-10-23; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- temozolomide maintain therapeutic (Experimental): Lobaplatin combined with etoposide for first-line treatment of extensive stage small cell lung cancer,then clinical benefit patients for temozolomide maintain therapeutic.This study have only one arm which temozolomide maintain at dose of 150mg/m2 D1-5 Q4W.
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: temozolomide — temozolomide maintain therapeutic
  Other Names: Temozolomide Capsule

SUMMARY:
This study evaluates temozolomide maintain therapeutic efficacy and safety in extensive stage SCLC who has clinical benefit from etoposide combined Los platinum (EL) scheme in the first line treatment.

DETAILED DESCRIPTION:
According to the etoposide combined Los platinum (EL) plan administration, every cycle was 21 days, a total of four cycle. The patients who was clinical benefit directly from EL scheme in the first line treatment accept temozolomide maintenance therapy, 150mg / m2, oral D1-5. A period of 28 days, regular follow-up and evaluation of effectiveness, safety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 70 years old, men and women are not limited;
2. confirmed by histopathological examination SCLC;
3. clinical stage for patients with extensive stage (except for the case of pleural effusion)
4. patients has no drug treatment history
5. the implementation of palliative radiotherapy for metastatic lesions, surgical treatment, after the end of treatment over 14 days.
6. there can be measured lesions (non radiation exposure site) of patients (RECIST) evaluation;
7. physical condition score ECOG PS:0-1
8. more than expected survival time over 3 months

Exclusion Criteria:

1. the previous platinum compounds have a history of allergies;
2. active ulcer patients;
3. Patients with primary lung lesions were treated with radiotherapy;
4. chest X-ray showed clear interstitial pneumonia or patients with pulmonary fibrosis;
5. the need for treatment of brain metastases in the active phase
6. there are more serious tumor invasion, superior vena cava syndrome, or in the middle volume of malignant pleural effusion, abdominal effusion or pericardial effusion, not yet control;
7. there is a serious infection, ADH abnormal secretion syndrome, poor control of diabetes,the need for the treatment of patients with severe complications such as vena cava syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival in the first line of chemotherapy | 6 months
  The first day of treatment to the date that disease progression is reported

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  The first day of treatment to death or last survival confirm date
Tumor Response Rate (RR) | 3 months
  The ratio between the number of responders and number of patients assessable for tumor response.
Treatment-related adverse events | the first date of treatment to 30 days after the last dose of study drug, assessed up to 6 months
  Treatment-related adverse events are assessed by common terminology criteria for adverse events (CTCAE) V4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No